CLINICAL TRIAL: NCT05966584
Title: RETENTION: An Open-Label Phase 2 Trial of InteRlEukin (5) InhibiTion for the prEveNTION of Alpelisib Rash in Metastatic PIK3CA-mutant Hormone-Receptor Positive Breast Cancer
Brief Title: A Study to Prevent Rash in People Starting Alpelisib for the Treatment of Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Limited amount of eligible participants
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: AstraZeneca (Industry); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-276
Record Dates: First submitted 2023-07-20; First posted 2023-07-28 (Actual); Results first posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer
Keywords: Alpelisib; Benralizumab; Metastatic HR-positive; HER2-negative breast cancer; Rash; 22-276
MeSH Terms: conditions — Breast Neoplasms; Exanthema | interventions — benralizumab; Fulvestrant; Alpelisib

STUDY DESIGN:
Intervention Model Description: A multi-center, open-label, phase 2 trial
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Benralizumab and PI3K inhibition (alpelisib) (Experimental): Patients will receive fulvestrant or AIs and PI3K inhibition (alpelisib) per SOC (fulvestrant on days 1, 15, 29 and monthly thereafter; Ais on a daily continuous basis). Participants will receive one injection of benralizumab 30mg subcutaneously on day -1.
  Interventions: Drug: Benralizumab; Drug: fulvestrant or AIs) and PI3K inhibition (alpelisib)

INTERVENTIONS:
Drug: Benralizumab — Benralizumab 30mg subcutaneously on day -1.
Drug: fulvestrant or AIs) and PI3K inhibition (alpelisib) — SOC endocrine therapy (fulvestrant or AIs) and PI3K inhibition (alpelisib)

SUMMARY:
The researcher are doing this study to find out whether benralizumab is effective at preventing skin rashes caused by alpelisib in people who have metastatic breast cancer. Skin rash is a common side effect of alpelisib. Researchers think adding benralizumab to the standard-of-care hormone treatment and alpelisib may prevent the patient from getting a rash.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic HR-positive, HER2-negative breast cancer. HR positive is defined by ER status >10% immunohistochemical (IHC) staining of any intensity.
2. Must be scheduled to receive SOC endocrine therapy (alpelisib plus fulvestrant or AIs)
3. Presence of one or more activating PIK3CA mutations in tumor tissue.
4. Measurable disease per RECIST v1.1 OR at least one predominantly lytic bone lesion must be present.
5. Written informed consent provided
6. Female or male ≥18 years of age
7. Eastern Cooperative Oncology Group performance status of 0 or 1.
8. Life expectancy ≥6 months.
9. Adequate organ and marrow function as defined below:

   * Hemoglobin ≥8.0 g/dL (without blood transfusion within 7 days of laboratory test used to determine eligibility)
   * Absolute neutrophil count ≥1.0 × 10^9 /L (without granulocyte colony stimulating factor support within 2 weeks of laboratory test used to determine eligibility)
   * Platelet count ≥50 × 10^9 /L (without transfusion within 2 weeks of laboratory test used to determine eligibility)
   * Total bilirubin (TB) ≤1.0 × institutional upper limit of normal (ULN; Patients with known Gilbert's disease who have TB ≤3 × ULN may be enrolled)
   * Aspartate transaminase/alanine transaminase ≤2.5 × ULN with normal alkaline phosphatase (≤5 × ULN for patients with liver metastases) OR ≤1.5 × ULN in conjunction with alkaline phosphatase >2.5 × ULN
   * Creatinine ≤1.5 mg/dL
10. Able to swallow oral medication.
11. Willing to be randomized to any of the treatment arms and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
12. Women must be of postmenopausal status. Postmenopausal status is defined by any one of the following criteria:

    * Prior bilateral oophorectomy
    * Age ≥60 years
    * Age <60 years and amenorrheic for at least 12 months (spontaneous cessation of menses for 12 consecutive months or more in the absence of chemotherapy, tamoxifen, toremifene, or ovarian suppression) and follicle-stimulating hormone and estradiol levels in the postmenopausal range without an alternative cause.

Exclusion Criteria:

1. Known hypersensitivity to alpelisib, fulvestrant or AIs, benralizumab, cetirizine, or to any of the excipients of alpelisib, fulvestrant or AIs, benralizumab, or cetirizine.
2. Concurrent malignancy (basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or cervical cancer in situ that have undergone curative intent therapy are allowed)
3. Individuals with impaired decision making capacity.
4. Concurrent use of another investigational drug or device for the rash (i.e., outside of study treatment) during, or within 4 weeks of treatment.
5. Known use of anti-IL-5 agents or other biologics for the treatment of asthma which are known to decrease blood eosinophil levels within the past 12 weeks.
6. Known history of anaphylaxis to benralizumab therapy.
7. A helminthic parasitic infection diagnosed within 24 weeks prior to the first treatment, and assent when applicable, was obtained that had not been treated with, or has failed to respond to, standard of care therapy.
8. Known history of human immunodeficiency virus (HIV) infection or current chronic or active hepatitis B or C infection requiring treatment with antiviral therapy.
9. Active infection that would impair the ability of the patient to receive study treatment.
10. Women who are pregnant or breast-feeding.
11. Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation.
12. Oral corticosteroids at a dose of ≥20mg/day prednisone or equivalent within 14 days expected to continue during alpelisib therapy.
13. More than 2 lines of endocrine-based therapy in the metastatic setting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-07-06 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2024-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alina Markova, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Rockville (Limited Protocol Activities), Rockville Centre, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Benralizumab and PI3K Inhibition (Alpelisib)
Started | 1
Completed | 0
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Benralizumab and PI3K Inhibition (Alpelisib)
Number analyzed (Participants) | 1
Age, Continuous [Mean (Full Range); unit: years] | 70 [70 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects That Have a Grade ≤1 Rash
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab and PI3K Inhibition (Alpelisib)
Number analyzed (Participants) | 1
Participants | 0

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Benralizumab and PI3K Inhibition (Alpelisib)
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-01): https://cdn.clinicaltrials.gov/large-docs/84/NCT05966584/Prot_SAP_000.pdf